CLINICAL TRIAL: NCT07207486
Title: In-depth Analysis of Cholesterol Metabolism and Related Biomarkers in the Pathogenesis and Progression of the Disease in Neurodegenerative Dementias
Acronym: RF-2021-123742
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: Università di Torino, Torino (Unknown); Ospedale San Luigi Gonzaga, Orbassano (Unknown)
Responsible Party: Sponsor
Other Study IDs: RF-2021-12374277
Record Dates: First submitted 2025-09-26; First posted 2025-10-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-09

CONDITIONS: Dementias; Neurodegenerative Dementia
Keywords: Cholesterol metabolism; Neurodegenerative dementias
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- AD: Patient with Alzheimer's disease
- FTD: Patient wirh Frontotemporal dementia
- PSP/CBD: Patient with tauopathy
- CN: Controll subjects

SUMMARY:
The aim of the study is to evaluate the role of cholesterol in the pathogenesis of neurodegenerative dementias. Hypercholesterolemia is a known risk factor for Alzheimer disease (AD), and oxysterols, the principal cholesterol metabolites, are involved in neuroinflammation, amyloid aggregation, and tau accumulation.

Oxysterols will be measured in different biological samples (post-mortem brain tissue, CSF, and plasma) from patients with different neurodegenerative dementias, including AD, frontotemporal dementia (FTD), and primary tauopathies. This approach will allow determination of whether their modifications correlate primarily with Aß deposition, tauopathy, or neuronal loss, with the goal of identifying correlations with disease severity and progression.

Since preliminary results suggest that the levels of most oxysterols in the brain significantly increase in parallel with the levels of the enzyme PCSK9, the investigators will explore the role of cholesterol metabolism and PCSK9 in AD and other dementias to evaluate whether cholesterol dysregulation represents a common alteration across these neurodegenerative disorders or is specific to AD

DETAILED DESCRIPTION:
The project is a monocentric retrospective and prospective low-intervention clinical study. All samples collected will be sent for analysis to the Laboratory of General Pathology and Pathophysiology, Department of Clinical and Biological Sciences, University of Turin, San Luigi Gonzaga Hospital, Orbassano (TO), Italy.

1. Selection and characterization of post-mortem brains Twenty brains from patients with AD (ranging from Braak stage II to VI of neurofibrillary pathology severity), ten brains from patients with FTD/tauopathies, and six brains from FTD/TDP43 patients will be included in the study. These samples are already available for the project and have been neuropathologically characterized by Neurology 5 - Neuropathology Unit.
2. Recruitment and follow-up of patients with neurodegenerative dementias

   Retrospective study Samples (CSF and plasma) previously collected from patients at Neurology 5 - Neuropathology Unit over the years will be used. The study will include 40 AD patients, 40 FTD patients, and 20 age-matched non-demented controls. Clinical and MRI data will be retrospectively collected, as well as levels of markers of neurodegeneration (tau, Abeta42, and phospho-tau) in CSF.

   Longitudinal study During the first 18 months of the project, 30 AD patients, 20 FTD patients, and 10 patients with primary tauopathies (PSP/CBD) will be recruited. A group of 20 age-matched healthy subjects will serve as controls. All patients and controls will undergo a comprehensive neurologic assessment, a neuropsychological evaluation, and a brain MRI with a standard protocol at baseline (T0) and after 1 year (T1). CSF collection will be performed at baseline in patients. DNA and plasma will be collected from controls and patients at baseline and follow-up. Measurements of BMI, total cholesterol, LDL and HDL cholesterol, and triglycerides will be performed at baseline and follow-up in all subjects. ApoE genotype will be analyzed for all subjects to determine E2, E3, and E4 polymorphisms. MRI will be performed on a 3T scanner, including volumetric T1, FLAIR, T2, DWI, and DTI sequences at baseline and follow-up.
3. Study of the role of the enzyme PCSK9 in the brain (performed by University of Turin) SK-N-BE cells and mouse-derived primary cortical neurons and astrocytes will be treated with PCSK9 or with an oxysterol mixture obtained from brain dosages.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-85
* Diagnosis based on the current diagnostic criteria for AD (McKhann et al., 2011), FTD (Gorno-Tempini et al., 2011; Rascovsky et al., 2011), PSP and CBD (Amstrong et al., 2013; Höglinger et al., 2017)
* Mini Mental State Examination MMSE > 10.

Exclusion Criteria:

* Other neurological or psychiatric disorders Severe chronic metabolic diseases

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will use samples (CSF and plasma) already collected from patients from Unit 1 over years. We will include 40 AD, 40 FTD and 20 age-matched non demented controls. Clinical and MRI data will be retrospectively collected as well as the levels of markers of neurodegeneration (tau, Abeta42 and phospho-tau) on CSF.
  Longitudinal study We will recruit 30 AD patients, 20 FTD patients and 10 patients with primary tauopathies (PSP/CBD) from out and inpatients of Neurology 5-Neuropathology Unit. A group of 20 age-matched subjects without neurological and/or psychiatric diseases will be enrolled as controls. The duration of enrolment will be 18 months.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2027-04-29 (Estimated); Study Completion 2027-04-29 (Estimated)

PRIMARY OUTCOMES:
Characterize differences in cholesterol precursors | 12 months
  To identify and characterize differences in cholesterol precursors and metabolites between patients with neurodegenerative dementias vs controls and between patients with different types of neurodegenerative dementia.

SECONDARY OUTCOMES:
different brain areas | 12 months
  To identify and characterize different levels of cholesterol precursors and metabolites as well as lipidomics and metabolomics changes in different brain areas of the same patients categorized as involved or spared by the different types of pathological changes.
cerebral oxysterol changes in AD | 12 months
  To find out whether cerebral oxysterol changes in AD (see preliminary results) involve globally the brain suggesting a general derangement of cerebral cholesterol metabolism or selectively brain areas involved by specific primary (Abeta deposition, tauopathy) or secondary (astrogliosis, microglial activation, neuroinflammation) alterations
different cholesterol precursors in neurodegenerative diseases examined in CSF and plasma | 12 months
  To identify different levels of cholesterol precursors and metabolites as well as lipidomics and metabolomics changes at different stages of the different neurodegenerative diseases examined in CSF and plasma.
cortical atrophy | 12 months
  To ascertain whether correlations exist between cholesterol precursors and metabolites abnormalities, severity of the disease, cortical atrophy, glial and microglial reactive changes and neuroinflammation in neurodegenerative dementias.
PCSK9 | 12 months
  To verify whether changes in the levels of PCSK9 and other cholesterol metabolism-related proteins are present in patients with the neurodegenerative dementias (brain tissue, CSF, and plasma).
PCSK9 in neurons | 12 months
  Levels of inflammatory markers and neurodegeneration-related proteins in neurons and astrocytes after treatment with PCSK9 in vitro.
potential neurotoxic action of PCSK9 | 12 months
  Efficacy of the new nanoparticle (NPs) formulation carrying anti-PCSK9 antibody in reducing PCSK9-induced neurotoxicity in neuronal and astrocyte cultures in vitro.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Università di Torino AOU San Luigi Gonzaga, Torino, to
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan

IPD SHARING:
Plan to Share IPD: No